CLINICAL TRIAL: NCT02055261
Title: Effects of Low Frequency Deep Brain Stimulation of the Pedunculopontine Nucleus on Gait and Balance Disorders of Parkinson's Disease
Brief Title: Pedunculopontine Nucleus Stimulation for Gait Disorders in Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pitié-Salpêtrière Hospital (Other)
Responsible Party: Principal Investigator, David Grabli, MD PhD, Pitié-Salpêtrière Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RBM C08-07
Record Dates: First submitted 2014-01-16; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFF PPN DBS-ON PPN DBS (Other): Patients randomly allocated to the order OFF Low frequency DBS of the pedunculopontine nucleus then ON Low frequency DBS of the pedunculopontine nucleus
  Interventions: Device: Low frequency DBS of the pedunculopontine nucleus
- ON PPN DBS - OFF PPN DBS (Other): Patients randomly allocated to the order ON Low frequency DBS of the pedunculopontine nucleus then OFF Low frequency DBS of the pedunculopontine nucleus
  Interventions: Device: Low frequency DBS of the pedunculopontine nucleus

INTERVENTIONS:
Device: Low frequency DBS of the pedunculopontine nucleus

SUMMARY:
The appearance of postural instability and gait disorders is a major turning point in the evolution of Parkinson's disease (PD). These axial symptoms are usually unresponsive to L-Dopa and represent a severe impairment for the patients due to frequent falls and reduced outside mobility. There is no effective pharmacological treatment available for these symptoms, and their pathophysiology is not well known : it is currently assumed that non-dopaminergic brainstem lesions participate to axial symptoms in PD. Surgically, these patients cannot benefit from high frequency deep brain stimulation (DBS) of the subthalamic nucleus (STN) since this operation tends to even aggravate axial symptoms unresponsive to L-Dopa in some patients. A dysfunction of the pedunculopontine nucleus (PPN) might be at the origin of these axial symptoms, since the PPN participates in the maintenance of posture and motion in primates. In PD patients, recent reports have suggested that low frequency stimulation of the PPN may equally improve gait and posture. However, these results are debatable due to methodological limitations, insufficient clinical evaluation and uncertain anatomical targeting. Thus, our aim is to propose a low frequency PPN stimulation to six advanced PD patients according to the usual criteria for STN DBS who are, however, unsuitable for this operation due to gait and posture disorders. We will perform a randomized, double-blind and cross over design (two months periods with and without DBS randomly assigned to each patient). The targeting will be allowed by a a three-dimensional and deformable atlas of the basal ganglia fusioned with the stereotaxic magnetic resonance imaging (MRI) of each patient. Evaluations will comprise 1 month before surgery and in "Off" and "On" stimulation condition:

* clinical motor assessment in both "Off" and "On" drug state, including cardinal parkinsonian signs, gait and balance
* gait initiation physiological evaluation
* cognitive and behavioral testing If our hypothesis is confirmed, low frequency PPN stimulation may well represent a substantial improvement of our therapeutic options for advanced PD patients suffering from debilitating gait and posture disorders unresponsive to L-Dopa.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Age < 70 and > = 18 years
* Improvement > or = 50 % during acute levodopa test
* Score > or = 2 on item 29 of UPDRS part 3 score obtained in "off" drug state
* No previous DBS
* No evidence of atypical parkinsonism
* No dementia (MATTIS > 129)
* No psychiatric disease
* Contraception if woman
* Informed consent

Exclusion Criteria:

* Contra indication to surgery
* Contra indication to MRI
* Severe life threatening comorbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change of Rating scale for gait evaluation between 'Off stim off drug" and "On stim off drug" conditions | 4 months and 6 months after surgery
  The primary outcome criteria will be the comparison between RSGE total score in obtained 'Off' and 'On' stimulation conditions either at 4 or 6 months after surgery according to the randomized order of the cross-over

SECONDARY OUTCOMES:
Adverse events records | 1 month before surgery, 1-2-3-4-5-6 months after surgery
Change of UPDRS part 3 score between "Off Stim Off drug" and "ON stim Off drug" conditions | 4 and 6 months after surgery
Change of Rating scale for gait evaluation between 'Off stim on drug" and "On stim on drug" conditions | 4 and 6 months after surgery
Change of UPDRS part 3 score between "Off Stim On drug" and "ON stim On drug" conditions | 4 and 6 months after surgery
Change of UPDRS part 3 score between "Off Stim Off drug" and "No stim Off drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of UPDRS part 3 score between "Off Stim On drug" and "No stim On drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of Rating scale for gait evaluation between 'Off stim Off drug" and "No stim off drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of Rating scale for gait evaluation between 'Off stim On drug" and "No stim on drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of Rating scale for gait evaluation between 'On stim Off drug" and "No stim off drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of Rating scale for gait evaluation between 'On stim On drug" and "No stim On drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of gait physiological parameters between "Off Stim Off drug" and "ON stim Off drug" conditions | 4 and 6 months after surgery
Change of gait physiological parameters between "Off Stim On drug" and "ON stim On drug" conditions | 4 and 6 months after surgery
Change of gait physiological parameters between "No Stim On drug" and "Off stim On drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of gait physiological parameters between "No Stim Off drug" and "On stim off drug" conditions | 1 month before surgery and 4 or 6 months after surgery
Change of gait physiological parameters between "No Stim Off drug" and "Off stim off drug" conditions | 1 month before surgery and 4 or 6 months after surgery

OTHER OUTCOMES:
Changes in sleep architecture between "off stim" and "on stim" conditions | 4 and 6 months after surgery
changes in cognitive evaluation between "Off stim" and 'On stim" conditions | 4 and 6 months after surgery
changes in cognitive evaluation between "No stim" and 'Off stim" conditions | 1 month before surgery and 4 or 6 months after surgery
changes in cognitive evaluation between "No stim" and 'On stim" conditions | 1 month before surgery and 4 or 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Pitié-Salpétrière, Paris, France